CLINICAL TRIAL: NCT04273932
Title: Effects of Lithium Therapy on Blood-based Therapeutic Targets in Parkinson's Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Professor of Neurology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003688
Record Dates: First submitted 2019-10-31; First posted 2020-02-18 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Lithium; Alpha-synuclein
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Lithium

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lithium aspartate 15mg a day (Experimental): 15mg of elemental lithium administered every morning by mouth.
  Interventions: Drug: Lithium
- Lithium aspartate 45mg a day (Experimental): 20mg every morning and 25mg every evening of elemental lithium administered by mouth.
  Interventions: Drug: Lithium
- Lithium carbonate (Experimental): The dose will be titrated based on weekly blood tests to achieve a target serum level of 0.40-0.50mmol/L, which represents an elemental lithium dose of about 85-170mg a day.
  Interventions: Drug: Lithium
- No lithium treatment (No Intervention): Control arm

INTERVENTIONS:
Drug: Lithium — Lithium aspartate of lithium carbonate will be administered by mouth.
  Arms: Lithium aspartate 15mg a day; Lithium aspartate 45mg a day; Lithium carbonate

SUMMARY:
This study aims to determine if one of three low doses of lithium therapy for 6 months can engage one or more blood-based therapeutic targets implicated in Parkinson's disease (PD) pathophysiology. Results of this study will help to determine if lithium therapy is worthwhile to further investigate as a potential disease-modifying therapy in PD, the optimal dose to study and the optimal PD subgroup most likely to benefit from lithium therapy.

DETAILED DESCRIPTION:
Lithium belongs to a class of kinase-targeting therapies, including the diabetes medication exenatide and the cancer medication nilotinib, that have demonstrated promise as disease-modifying therapies for Parkinson's disease (PD). Exenatide was recently shown to engage protein kinase B (Akt) and provide significant symptomatic and possible disease-modifying benefit in PD in a phase 2 randomized controlled trial (RCT). Nilotinib engages c-Abelson kinase (c-Abl) and its disease-modifying effects are currently being investigated in two, phase 2 PD RCTs. Lithium targets Akt, glycogen synthase kinase-3 beta (GSK-3B, a downstream target of Akt) and cyclin-dependent kinase 5 (cdk5, a downstream target of c-Abl) in manners that recapitulate those of exenatide and nilotinib. Also, lithium inhibits inositol monophosphate leading to enhanced autophagy and reduced intracellular levels of alpha-synuclein (a-synuclein), which is believed to be a primary mediator of the progressive neurodegeneration in PD. In addition to a-synuclein, genome-wide association studies (GWAS) have implicated oligomeric tau in the pathogenesis of PD. Pathological mutations in leucine-rich repeat kinase 2 (LRRK2) are the most common genetic cause of a late-onset parkinsonism that is clinically indistinguishable from sporadic PD and very similar pathologically. Pathological LRRK2 mutations affect the activities of Akt, GSK-3B and cdk5 to greatly increase the formation of phosphorylated tau (p-tau) - the precursor to tau oligomer formation - and decrease the activity of the transcriptional cofactor B-catenin - which mediates the transcription of neuronal survival genes implicated in PD such as nuclear receptor related 1 (Nurr1). Through its ability to inhibit GSK-3B, lithium can enhance B-catenin-mediated activity and Nurr1 expression. Lithium was also effective in several PD animal models. Finally, both clinical trial and epidemiologic data suggest that lithium exposures of even <1mg a day may provide significant disease-modifying effects in neurodegenerative diseases including PD.

The investigators propose to assess the effects of 3 lithium dosages for 6 months on the above targets measured in blood in a randomized, parallel design, proof of concept clinical trial among 18 PD patients. In addition, 2 PD patients will serve as controls and not receive lithium therapy.

ELIGIBILITY:
1. Diagnosed with PD according to the UK Brain Bank Criteria.
2. 45-80yo.
3. Clinical Dementia Rating Scale score of 0 or 0.5.
4. Stable PD medications for previous 30 days and no current need for changes in the opinion of the PI.
5. No formed visual hallucinations or delusions for previous year.
6. Never taken prescription or over-the-counter lithium.
7. Stable or no diuretics for past 4 weeks and no need for changes for at least 6 months, in the PI's opinion.
8. Stable doses of antidepressants, antihypertensives and non-steroidal anti-inflammatory medications (NSAIDs) for previous 60 days and no current need to adjust such medications.
9. No history of cardiac arrhythmias besides atrial fibrillation that is rate controlled.
10. No unstable cardiac, medical or psychiatric condition in the opinion of the PI.
11. No current use of illicit drugs or current alcohol abuse in the opinion of the PI.
12. No history of hypothyroidism, not receiving thyroid replacement therapy and normal thyroid stimulating hormone (TSH) level at screening visit.
13. Estimated renal glomerular filtration rate ≥50 at screening visit.
14. No history of receiving or planning to receive nilotinib or a glucagon-like peptide-1 agonist medication such as exenatide.
15. No use of tobacco products for the previous year.
16. No deep brain stimulation (DBS) or possible need for DBS for at least 1-year in the opinion of the PI.
17. Women with child bearing potential will need a negative pregnancy test and not be nursing an infant at screening. Women with child bearing potential will need to report using barrier method or hormonal contraception.
18. Not enrolled in another clinical trial.
19. Willing and able to sign informed consent and follow study procedures.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Plasma alpha-synuclein assessed by ultra-sensitive, immunomagnetic reduction assay (MagQu, LLC, Surprise, AZ). | Change from baseline to 24 weeks
Peripheral blood mononuclear cell (PBMC) Nurr1 mRNA levels by real-time polymerase chain reaction. | Change from baseline to 24 weeks
PBMC phosphorylated (p) and total (t) levels of pSerine9 and t-glycogen synthase kinase-3B | Change from baseline to 24 weeks
Plasma brain-derived neurotrophic factor (BDNF). | Change from baseline to 24 weeks
PBMC pThreonine308 and t-protein kinase B (Akt). | Change from baseline to 24 weeks

SECONDARY OUTCOMES:
Trough, steady-state plasma lithium levels by ICP/MS | Change from baseline to 24 weeks
Patient tolerability | Up to 24 weeks
  Assessed by patient reported adverse events.
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III (Motor Examination) and question 1.11 (Constipation Problems) in the "on" state | Change from baseline to weeks 12 and 24.
  Score range 0-132 with higher values indicating more severe symptoms.
Parkinson's Anxiety Scale | Change from baseline to weeks 12 and 24.
  Score range 0-48 with higher values indicating more severe symptoms.
Geriatric Depression Scale-15 | Change from baseline to weeks 12 and 24.
  Score range 0-15 with higher values indicating more severe symptoms.
Fatigue Severity Scale | Change from baseline to weeks 12 and 24.
  Score range 9-56 with higher values indicating more severe symptoms.
Insomnia Severity Index | Change from baseline to weeks 12 and 24.
  Score range 0-28 with higher values indicating more severe symptoms.
Parkinson's Disease Questionnaire-8 | Change from baseline to weeks 12 and 24.
  Score range 0-32 with higher values indicating more severe symptoms.
Montreal Cognitive Assessment (MoCA) | Change from screening to week 24
  Score range 0-30 with higher values indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Williamsville, New York, United States

REFERENCES:
- [Result] Guttuso T Jr, Shepherd R, Frick L, Feltri ML, Frerichs V, Ramanathan M, Zivadinov R, Bergsland N. Lithium's effects on therapeutic targets and MRI biomarkers in Parkinson's disease: A pilot clinical trial. IBRO Neurosci Rep. 2023 May 7;14:429-434. doi: 10.1016/j.ibneur.2023.05.001. eCollection 2023 Jun. PMID 37215748
- See also: PubMed Link to study results — http://www.ncbi.nlm.nih.gov/pubmed/37215748